CLINICAL TRIAL: NCT01441349
Title: A Randomized Phase II Study of Irinotecan/Cisplatin With or Without Simvastatin in Chemo-naive Patients With Extensive Disease-small Cell Lung Cancer
Brief Title: Irinotecan/Cisplatin With or Without Simvastatin in Chemo-naive Patients With Extensive Disease-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ji-youn Han, Head, lung cancer center, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-11-527
Record Dates: First submitted 2011-09-14; First posted 2011-09-27 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Simvastatin; SCLC; Extensive Disease
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Active Comparator): IP chemotherapy arm
  Interventions: Drug: IP chemotherapy
- Treatment arm (Experimental): IP chemotherapy plus simvastatin arm
  Interventions: Drug: IP chemotherapy plus simvastatin

INTERVENTIONS:
Drug: IP chemotherapy — Irinotecan/cisplatin (IP) chemotherapy
  * Cisplatin(30 mg/m2) diluted into 150 ml of 0.9% NS for IV over 30 min on day 1 &8.
  * Irinotecan(65mg/m2) diluted into 200ml of 5DW IV over 90 min on day 1 & 8
  * Every 21 days
  Other Names: IP
  Arms: Control arm
Drug: IP chemotherapy plus simvastatin — * Cisplatin(30mg/m2)diluted into 150 ml of 0.9% NS for IV over 30 min on day 1 &8
  * Irinotecan( 65 mg/m2) diluted into 200ml of 5DW IV over 90 min on day 1& 8.
  * Every 21days.
  * Simvastatin 40 mg per day orally D1of cycle 1
  Other Names: IPSimva
  Arms: Treatment arm

SUMMARY:
The purpose of this study is to compare the efficacy of Simvastatin and Irinotecan/Cisplatin chemotherapy with Irinotecan/Cisplatin chemotherapy alone in Extensive disease-small cell lung cancer.

DETAILED DESCRIPTION:
Statins (3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors) have been used to treat hypercholesterolemia. Besides the lipid lowering effects, they also act as anti-inflammatory and anti-cancer agents. Recently the investigators demonstrated a synergistic cytotoxicity between Simvastatin and Irinotecan in human lung cancer cells. Simvastatin enhances Irinotecan-induced apoptosis by inhibition of proteasome activity. All of these additional actions may counteract harmful effects of smoking-induced chronic inflammation. These properties together with a high safety profile have made Statins more attractive drug for small cell lung cancer (SCLC), the highly smoking-related cancer.

Given the promising preclinical anti-tumor and anti-inflammatory effects of Simvastatin in SCLC, recently the investigators conducted a phase II study of Simvastatin and Irinotecan/Cisplatin (IP) chemotherapy in chemo-naïve- patients with Extensive disease-small cell lung cancer (ED-SCLC). The 1-year survival rate was 39.3%. The median overall survival (OS) and progression free survival (PFS) was 11.0 months and 6.1 months, respectively. Overall relative risk (RR) was 75%. The most common toxicity was neutropenia (67%). The efficacy was significantly associated with smoking-status. Compared with never-smokers, ever-smokers had higher RR (40% v 78%, P=0.01) and longer PFS (2.5 months v 6.4 months, P=0.018) and showed a trend toward improved OS (9.0 months v 11.2 months, P=0.095). The effect of smoking on survival was apparent when subdividing ever smokers according to pack-years (PY). Ever-smokers who smoked > 65 PY showed significantly longer OS compared to ever-smokers who smoked <= 65 PY or never-smokers (20.6 months v 10.6 months v 9.0 months, log-rank P=0.032). In multivariate analysis, PY > 65 was predictive for longer survival (hazard ratio) HR=0.377 [95% CI (confidence interval), 0.157-0.905]). These findings suggest that the addition of Simvastatin to Irinotecan and Cisplatin improved efficacy in ever-smokers with ED-SCLC. The survival benefit of this combination seems apparent in heavy-smokers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed SCLC
* Extensive - stage disease, defined as disease extending beyond one hemithorax or involving contralateral mediastinal, hilar or supraclavicular lymph nodes, and/ or pleural effusion
* ever smoker( have smoked> 100 cigarettes in entire lifetime
* No prior chemotherapy, immunotherapy, or radiotherapy
* Measurable disease according to RECIST 1.1
* Patient compliance that allow adequate follow - up
* Adequate hematologic , hepatic and renal function.
* Written informed consent that is consistent with International Conference on Harmonization (ICH) - Good Clinical Practice (GCP) guidelines
* Males of females at least 18 years of age
* If female : childbearing potential either terminated by surgery, radiation, or menopause or attenuated by use of an approved contraceptive method(intrauterine device, birth control pills, or barrier device)during for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative hCG test within 7 days prior to the study enrollment.
* No concomitant prescriptions including cyclosporin A, valproic acid, phenobarbital, phenytoin, ketoconazole.
* Patients with brain metastasis are allowed unless there were clinically significant neurological symptoms or signs.

Exclusion Criteria:

* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction with 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Concurrent administration of any other antitumor therapy.
* Pregnant or Breast-feeding.
* Taking simvastatin or Any contraindications for therapy with simvastatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2011-08 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year survival rate | every 8 weeks
  Survival time will be calculated from the date of study treatment start to the date of death.( or date last seen ) Follow - up visits are conducted every 8 weeks to obtain meaningful data on time- to event variables. Assessment will continue until death or 12 months after treatment.

SECONDARY OUTCOMES:
Tumor Response rate | every 2 cycles or 6 weeks
  The response rate will be determined by the number of patients with complete and partial responses according to RECIST criteria 1.1
Progression free survival | every 2 cycles or 6 weeks.
  Progression free survival will be calculated from the date of study treatment start to the first objective documentation of progressive disease or to the date of death, whichever occurs first.
Toxicity profile | every 3 weeks
  Safety will be evaluated by the frequency, severity, and relationship of adverse event graded by NCI Common Toxicity Criteria version 4.0 that occur during the treatment and follow up periods.

CONTACTS AND LOCATIONS:
Overall Officials: JI-YOUN HAN, M.D. PhD., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center , Korea, Goyang-si, Gyeonggi-do, South Korea